CLINICAL TRIAL: NCT02388490
Title: A Phase II Study of Brentuximab Vedotin in Patients With Relapsed or Refractory EBV-and CD30-positive Lymphomas
Brief Title: Brentuximab Vedotin in Patients With Relapsed or Refractory EBV-and CD30-positive Lymphomas
Acronym: Bretuximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X25016
Record Dates: First submitted 2015-02-04; First posted 2015-03-17 (Estimated); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2019-04

CONDITIONS: Relapsed or Refractory EBV-and CD30-positive Lymphomas
Keywords: Brentuximab vedotin; EBV; Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brentuximab vedotin (Experimental): Brentuximab vedotin is an antibody-drug conjugate (ADC) composed of the anti-CD30 chimeric immunoglobulin G1 (IgG1) monoclonal antibody cAC10 and the potent antimicrotubule drug monomethyl auristatin E connected by a protease-cleavable linker. cAC10 binds to the CD30 antigen, which has a very low expression on normal cells but is found on some tumor cells.
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — Brentuximab vedotin administered by IV infusion given over approximately 30 minutes on Day 1 of each 21-day cycle. The dose of brentuximab vedotin is 1.8 mg/kg q 3 weeks.
  Other Names: Adcetris

SUMMARY:
This is an open-label, non-randomized, multi-center, phase II trial of brentuximab vedotin to evaluate ORR primarily in patients with EBV- and CD30-positive lymphomas.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, multi-center, phase II trial of brentuximab vedotin to evaluate ORR primarily in patients with EBV- and CD30-positive lymphomas. The ORR will be evaluated based on the revised Cheson's criteria or modified SWAT criteria in case of cutaneous EBV- and CD30-positive lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory EBV- and CD30-positive lymphomas
2. Age ≥ 18 years
3. ECOG performance status 0-2
4. At least one measurable lesion based on revised Cheson's or modified SWAT criteria
5. Provision archival tumor tissues (4 μm thickness x 5 unstained slides) and blood samples
6. Voluntary written informed consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
7. Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
8. Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
9. Adequate hematologic function: absolute neutrophil count (ANC) ≥1,500/µL, platelet count ≥ 75,000/µL, and hemoglobin ≥8.0 g/dL unless there is known hematologic tumor marrow involvement (ANC ≥ 1,000/µL and platelet count ≥ 50,000/µL if there is known bone marrow involvement)
10. Adequate liver function: total bilirubin < 1.5 x the upper limit of the normal (ULN) unless the elevation is known to be due to Gilbert syndrome and ALT or AST < 3 x ULN (AST and AST < 5 x ULN if their elevation can be reasonably ascribed to the presence of hematologic tumor in liver)
11. Adequate renal function: serum creatinine < 2.0 mg/dL and/or creatinine clearance or calculated creatinine clearance > 40 mL/minute.
12. Expected survival > 3 months

Exclusion Criteria:

1. Female patient who are both lactating and breast-feeding or have a positive serum pregnancy test
2. Any serious medical or psychiatric illness
3. Known cerebral or meningeal involvement (EBV- and CD30-positive lymphoma or any other etiology), including signs or symptoms of PML
4. Symptomatic neurologic disease compromising normal activities or requiring medication
5. Any sensory or motor peripheral neuropathy greater than or equal to Grade 2
6. Known history of myocardial infarction within 1 year, NYHA class III/IV heart failure, or uncontrolled cardiovascular conditions including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%.
7. Any active systemic viral, bacterial, or fungal infection within 2 weeks prior to first study drug dose
8. Any prior chemotherapy and/or other investigational agents within at least 5 half-lives of last dose
9. Prior stem cell transplantation within 100 days or radioimmunotherapy within 8 weeks
10. Prior exposure to CD30-targeted agents
11. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin
12. Known human immunodeficiency virus (HIV) positive
13. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
14. Another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae Min Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National Unversity Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul

REFERENCES:
- [Derived] Kim M, Lee JO, Koh J, Kim TM, Lee JY, Jeon YK, Keam B, Kim DW, Lee JS, Heo DS. A phase II study of brentuximab vedotin in patients with relapsed or refractory Epstein-Barr virus-positive and CD30-positive lymphomas. Haematologica. 2021 Aug 1;106(8):2277-2280. doi: 10.3324/haematol.2021.278301. No abstract available. PMID 33792222

RESULTS

PARTICIPANT FLOW:
Groups:
- Brentuximab Vedotin: This group was consisted of patients with EBV-positive and CD30- positive non-Hodgkin lymphomas with various levels of CD30 in the relapsed or refractory setting and designed to evaluate the activity of brentuximab vedotin in the patients.
  Brentuximab vedotin was administered by IV infusion, given over approximately 30 minutes on Day 1 of each 21-day cycle. The dose of brentuximab vedotin is 1.8 mg/kg, q 3 weeks.
Period: Overall Study
Arm/Group | Brentuximab Vedotin
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Brentuximab Vedotin: This group was consisted of patients with EBV-positive and CD30- positive non-Hodgkin lymphomas with various levels of CD30 in the relapsed or refractory setting and designed to evaluate the activity of brentuximab vedotin in the patients.
  Brentuximab vedotin: Brentuximab vedotin administered by IV infusion given over approximately 30 minutes on Day 1 of each 21-day cycle. The dose of brentuximab vedotin is 1.8 mg/kg q 3 weeks.
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 67 [38 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 25

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Overall Response Rate (ORR) of Brentuximab Vedotin in EBV- and CD30-positive Lymphomas
Description: The primary endpoint was the ORR based on the revised criteria or modified Severity Weighted Assessment Tool (SWAT) criteria in the case of cutaneous lymphomas.
Time Frame: One-year
Population: Revised tumor response criteria for lymphoma(Revised Cheson) or revised SWAT and assessed by MRI except a pregnant patient whose response evaluation can be assessed by CT scan: Complete Response (CR), Disappearance of all evidence of the disease; Partial Response (PR), Regression of measurable disease and no new lesions. The SPD of the largest 6 major nodules should decrease by ≥ 50%, and there should be no increase in the size of other nodules; Overall Response (OR) = CR + PR.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 25
Participants | 12

2. Secondary Outcome: To Evaluate the Safety Profile
Description: AEs/SAEs occurring during the study period defined by CTCAE version 4.03
Time Frame: From the first dose of brentuximab vedotin to up to 30 days after the last dose, a total of up to approximately 366 days
Population: Among 25 patients, treatment-related serious adverse reactions were observed in 9 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 25
Participants | 9

3. Secondary Outcome: To Calculate Progression-free Survival (PFS) Time
Description: PFS as defined as the time from the date of initiation until the date of first documented progression.
  Revised tumor response criteria for lymphoma(Revised Cheson) or revised SWAT and assessed by MRI except a pregnant patient whose response evaluation can be assessed by CT scan: Progression is defined using these criteria, as observation of a new lesion or an increase of 50% or more from the nadir in a previously involved site.
Time Frame: One-year
Population: Clinical outcomes of brentuximab vedotin treatment according to lymphoma subtype and CD30 expression.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 25
months
  All | 6.1 [2.8 to 13.5]
  Mature T/NK cell: number analyzed (Participants) | 22
  Mature T/NK cell | 6.1 [0 to 13.9]
  Mature B cell: number analyzed (Participants) | 3
  Mature B cell | 3.0 [0.5 to 5.5]
  CD 30 expression < 10%: number analyzed (Participants) | 13
  CD 30 expression < 10% | 5.5 [0 to 15.3]
  10% <= CD 30 expression < 50%: number analyzed (Participants) | 5
  10% <= CD 30 expression < 50% | 9.7 [0 to 24.3]
  50% <= CD 30 expression: number analyzed (Participants) | 7
  50% <= CD 30 expression | 6.1 [0 to 14.6]

4. Secondary Outcome: To Calculate the Duration of Response
Description: The duration of response was assessed in 12 patients who had objective responses. The response continued even after the completion of the planned 16 cycles of brentuximab vedotin administration in three of these 12 patients (25%) at the time of data cut-off.
Time Frame: From the first dose Up to the time of data cut-off.
Population: The duration of response was assessed in 12 patients who had objective responses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 12
months | 10 [4.2 to 21.0]

5. Secondary Outcome: To Calculate Overall Survival (OS) Time
Description: OS as defined as the time from the date of first dose until death due to any cause.
  The median overall survival was obtained, but the upper value of 95% Confidence Interval was not reached at the time of data cut-off. Therefore the longest OS was 30.4 months, the follow-up duration up to the date of data cut-off.
Time Frame: From first dose to end of data collection
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 25
months | 15.6 [6.1 to 30.4]

6. Other Pre Specified Outcome: The Number of Participants With a Tumor Response Stratified by CD30-positive Expression
Description: Exploratory. The level of soluble CD30 (sCD30) was determined using an enzyme-linked immunosorbent assay.
Time Frame: One-year
Population: The level of soluble CD30 (sCD30) was determined using an enzyme-linked immunosorbent assay.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 25
Participants
  CD30 expression < 10%: number analyzed (Participants) | 13
  CD30 expression < 10%: CR | 2
  CD30 expression < 10%: PR | 4
  CD30 expression < 10%: Non-CR and Non-PR | 7
  10% <= CD30 expression < 50%: number analyzed (Participants) | 5
  10% <= CD30 expression < 50%: CR | 3
  10% <= CD30 expression < 50%: PR | 0
  10% <= CD30 expression < 50%: Non-CR and Non-PR | 2
  50% <= CD30 expression: number analyzed (Participants) | 7
  50% <= CD30 expression: CR | 0
  50% <= CD30 expression: PR | 3
  50% <= CD30 expression: Non-CR and Non-PR | 4

7. Other Pre Specified Outcome: Exploratory.
Description: The level of soluble CD30 (sCD30) was determined using an enzyme-linked immunosorbent assay. The specimen were collected on the date of screening visit.
Time Frame: On the date of screening visit.
Population: The median value of soluble CD30 (sCD30) was obtained.
Measure: Median (95% Confidence Interval); unit: ng/mL
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 25
ng/mL | 99.03 [2.67 to 2155.78]

8. Other Pre Specified Outcome: The ORR in the Groups With High sCD30 (≥ 99.03 ng/mL) and Low sCD30 (<99.03 ng/mL).
Description: The ORR in the groups with high sCD30 (≥ 99.03 ng/mL) and low sCD30 (<99.03 ng/mL) were determined up to the date of data cut-off.
Time Frame: Up to the date of data cut-off
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 25
Participants
  The ORR in the groups with high sCD30 (1-<10%) | 13
  The ORR in the groups with intermediate sCD30 (10-<50%) | 5
  The ORR in the groups with low sCD30 (>=50%) | 7

ADVERSE EVENTS:
Time Frame: From the day of first IP administration to 30 days after the last IP administration(till PD or unacceptable toxicity), an average of 1 year
Arm/Group | Brentuximab Vedotin
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=25)
Fracture (Musculoskeletal and connective tissue disorders) | 1 — Fracture of femur neck
Herpes zoster (Skin and subcutaneous tissue disorders) | 3
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (Psychiatric disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Cytopenia (Blood and lymphatic system disorders) | 1 — Platelet count decreased
Neutropenia (Blood and lymphatic system disorders) | 1 — Neutrophil count decreased
Hematuria (Renal and urinary disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Fungal infection (Infections and infestations) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
General weakness (Endocrine disorders) | 1
Neck mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=25)
Peripheral neutropathy (Nervous system disorders) | 12
Neutropenia (Immune system disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3
Fatigue (Psychiatric disorders) | 3
Anemia (Blood and lymphatic system disorders) | 1
Decreased appetite (Psychiatric disorders) | 2
Pruitus (Skin and subcutaneous tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Hyperglycemia (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Asthenia (Nervous system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 1
Nail change (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Sore throat (Ear and labyrinth disorders) | 1
Thirst (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT02388490/Prot_SAP_000.pdf